CLINICAL TRIAL: NCT07182734
Title: Feasibility of Unsupervised Therapy After Neurological or Orthopaedical Injury in the Home Setting With a Hand Rehabilitation Device (ReHandyBot) and an Assistive Smartphone Application (RehabCoach): an Exploratory Study
Brief Title: Feasibility of Unsupervised Therapy After Neurological or Orthopaedical Injury in the Home Setting With a Hand Rehabilitation Device (ReHandyBot) and an Assistive Smartphone Application (RehabCoach)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Rehaklinik Bellikon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RHB Home - RehabCoach
Record Dates: First submitted 2025-09-03; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rehabilitation After Neurological or Orthopaedic Injuries
Keywords: rehabilitation; stroke; traumatic brain injury; robotic devices; unsupervised therapy; hand training; upper limb therapy
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReHandyBot + RehabCoach (neurological) (Experimental): Participants will use the ReHandyBot hand rehabilitation device together with the RehabCoach smartphone app. All participants will:
  * Complete a preparation phase with screening and baseline clinical assessments.
  * Perform 3 supervised 30-minute training sessions with ReHandyBot in the clinic.
  * Perform 3-7 minimally supervised 30-minute training sessions in the clinic, with daily use of RehabCoach.
  * If ready, continue into an unsupervised phase, taking ReHandyBot home for daily training (recommended at least 30 minutes per day), supported by RehabCoach.
  * Return for a final evaluation including clinical and robotic assessments and usability feedback.
  Interventions: Device: Supervised and minimally-supervised therapy with ReHandyBot and RehabCoach; Device: Unsupervised Therapy with ReHandyBot and RehabCoach
- ReHandyBot + RehabCoach (orthopaedic) (Experimental): Participants will use the ReHandyBot hand rehabilitation device together with the RehabCoach smartphone app. All participants will:
  * Complete a preparation phase with screening and baseline clinical assessments.
  * Perform 3 supervised 30-minute training sessions with ReHandyBot in the clinic.
  * Perform 3-7 minimally supervised 30-minute training sessions in the clinic, with daily use of RehabCoach.
  * If ready, continue into an unsupervised phase, taking ReHandyBot home for daily training (recommended at least 30 minutes per day), supported by RehabCoach.
  * Return for a final evaluation including clinical and robotic assessments and usability feedback.
  Interventions: Device: Supervised and minimally-supervised therapy with ReHandyBot and RehabCoach; Device: Unsupervised Therapy with ReHandyBot and RehabCoach

INTERVENTIONS:
Device: Supervised and minimally-supervised therapy with ReHandyBot and RehabCoach — During the familiarization phase at the rehabilitation clinic, participants perform one week of supervised and one week of minimally-supervised therapy with the ReHandyBot under the supervision of a therapist or researcher. Minimally-supervised therapy means that participants try to perform therapy independently with the device, while the supervisor is present to provide assistance only if problems occur or if participants have questions.
  A few days after the study begins, participants are introduced to the RehabCoach application, which provides conversational support, reminders, and educational content throughout the intervention.
  During the supervised and minimally-supervised phases (first 2 weeks), the intervention dose is 5 sessions of approximately 45 minutes per week. These sessions are performed in addition to the conventional therapy plan. In each session, the robot proposes a set of 3 exercises, each lasting between 10 and 15 minutes.
Device: Unsupervised Therapy with ReHandyBot and RehabCoach — After the familiarization phase, participants continue training without direct supervision at the clinic until discharge and then at home for six weeks. If the therapist considers the participant capable of training safely and effectively with the device, the participant will keep training with the ReHandyBot unsupervised, both at the clinic and at home, while supported by the RehabCoach application. RehabCoach provides reminders, motivational support, and educational material to guide the home-based therapy.
  If participants are not considered ready for unsupervised therapy with the device, they will not proceed to the unsupervised phase.

SUMMARY:
The goal of this clinical trial is to evaluate whether using the ReHandyBot hand rehabilitation device together with the RehabCoach smartphone app can support safe, independent, and effective home therapy in patients with stroke, traumatic brain injury, or orthopedic problems.

The main questions it aims to answer are:

* Can patients safely and independently use ReHandyBot and RehabCoach after leaving the clinic?
* Will patients follow the recommended daily therapy schedule when using these tools at home?
* How do patients experience the usability and acceptability of ReHandyBot and RehabCoach in everyday life?
* Can this type of home-based therapy be extended to populations beyond stroke, such as traumatic brain injury and orthopedic patients?

Participants will:

* Complete a screening and baseline assessment with a therapist.
* Use ReHandyBot in a supervised phase at the clinic (3 sessions of 30 minutes).
* Continue with a minimally supervised phase at the clinic (3-7 sessions of 30 minutes, with daily app use).
* If ready, enter the unsupervised phase, taking ReHandyBot home for daily 30-minute training sessions, supported by RehabCoach.
* Return for a final assessment including clinical and robotic evaluations and usability feedback.

DETAILED DESCRIPTION:
Many neurological (e.g., stroke, traumatic brain injury) and orthopedic patients do not fully recover hand function, with a consequent decrease in independence and quality of life. Growing evidence shows that increasing the dose of upper limb therapy for in- and outpatients could improve functional outcomes. However, due to limited resources such as the low number of therapists, providing a higher dose of therapy to patients after discharge is highly challenging.

Unsupervised technology-assisted therapy, i.e., patients training with rehabilitation technologies without external supervision or intervention, may allow an increase in therapy dose (in clinical settings and at home) with little impact on the additional resources needed.

At the Rehabilitation Engineering Laboratory (RELab, ETH Zurich) we developed ReHandyBot, a portable device for hand rehabilitation. ReHandyBot was developed for unsupervised application in the home setting and preliminary results of an ongoing study show that stroke patients can learn how to use the device independently and bring it home to keep training with it after discharge from the clinic, increasing their therapy dose. However, during the unsupervised phase at home, patients' adherence to the recommended dose of therapy with ReHandyBot (i.e., at least one therapy session per day) was not always optimal.

At home, without the supervision of healthcare providers, patients often experience a decline in motivation and engagement over time. To address this, we developed RehabCoach, a smartphone application designed to support unsupervised therapy with ReHandyBot. RehabCoach incorporates chatbots (i.e., conversations with virtual assistants) and gamification elements designed to enhance therapy adherence. Until now, RehabCoach has been tested in some pilot usability studies, but a more extended evaluation has not been performed yet.

This study, therefore, investigates the use of ReHandyBot supported by RehabCoach at the homes of patients with stroke, traumatic brain injury, or orthopedic issues. The main objectives of this study are therefore to investigate (i) the feasibility of unsupervised therapy with ReHandyBot and RehabCoach within patients' home after discharge from the clinic, (ii) compliance to the therapy schedule after discharge, (iii) the usability of ReHandyBot and RehabCoach and user experience when using them, and (iv) the feasibility of extending therapy with ReHandyBot to populations other than stroke (i.e., patients with orthopedic problems or traumatic brain injury).

Sex and gender are not relevant for this study, as we do not expect the feasibility of using the device without supervision to be dependent on them.

The primary objective of this study is to investigate feasibility of unsupervised home therapy with the ReHandyBot supported by RehabCoach and to determine subjects' compliance to unsupervised robot-assisted therapy in the home setting as measured by the amount of self-administered dose of therapy with ReHandyBot.

Main secondary objectives comprise the evaluation of usability of ReHandyBot and RehabCoach and of user experience during robot-assisted therapy and when using the app, the feasibility of extending therapy with ReHandyBot to individuals with traumatic brain injury or orthopedic injury, functional recovery of the upper limb, parameters possibly influencing the use of ReHandyBot and RehabCoach, the impact of the goal and reward systems implemented on RehabCoach on motivation to train with ReHandyBot, as well as the feasibility and usability of the educational program delivered by the app.

The primary outcome of this study is the dose (e.g., therapy time, number of repetitions) of self-administered robot-assisted therapy performed by subjects in the home setting without supervision.

Main secondary outcomes are the number of subjects who can use ReHandyBot and RehabCoach unsupervised at home out of the total number of tested subjects, attendance to the therapy schedule during the unsupervised phase at home, adherence to the interactions required by RehabCoach, the number of times and reasons why the investigators need to intervene to help participants with eventual issues during the phase at home, safety, usability of ReHandyBot and RehabCoach and user experience (System Usability Scale, mHealth App Usability Questionnaire for RehabCoach, Customer Satisfaction Score, Net Promoter Score, open interview, etc.), number of additional therapy sessions initiated by the patients compared to the minimum recommendations, functional recovery.

Participants will receive robot-assisted therapy sessions with the ReHandyBot in parallel to their conventional therapy program for a period of around nine weeks. Additionally, they will interact with an app, RehabCoach, which will motivate patients to maximize the amount of training they perform with ReHandyBot.

This study consists of the following phases:

* Preparation phase: This phase includes a screening visit and an evaluation session with a therapist to perform baseline clinical assessments.
* Supervised phase: During the first week, subjects perform 3 sessions of 30 minutes of therapy with ReHandyBot supervised by a therapist or researcher. This phase is performed at the clinic and is used to familiarize the subject with the rehabilitation device. Additionally, the participants are also introduced to RehabCoach.
* Minimally supervised phase: During the second week, subjects interact with RehabCoach daily and perform 3-7 sessions of 30 minutes of minimally supervised therapy with the device at the clinic. The supervisor is still present but helps only in case patients encounter problems or if they have any questions. At the end of this phase, the supervisor uses a checklist to determine if the subject can proceed to the unsupervised phase. If not, the participant stops the study at the end of the minimally supervised phase. At the end of the minimally supervised phase, subjects need to fill in some questionnaires to rate the usability of ReHandyBot and RehabCoach.
* Unsupervised phase: If patients are ready for unsupervised training, during the unsupervised phase they take the ReHandyBot home and have the opportunity to independently exercise with the robot, with the recommendation of training at least 30 minutes per day (i.e., one complete therapy session per day) but also informing them that the more they train, the better. Patients who can use RehabCoach at home will also continue with the daily interactions with the app.
* Final phase: At the end of the protocol, subjects repeat the clinical and robotic assessments and the usability evaluation.

ELIGIBILITY:
Eligibility criteria for neurological patients

Inclusion criteria:

* Informed Consent signed by the subject.
* Female and male patients between 18 and 90 years old.
* Stroke or traumatic brain injury (recruitment within 6 months from event onset).
* Presence of a motor and/or sensory impairment of the upper limb as assessed by the responsible therapist.
* Possibility (e.g., enough space) to set up the ReHandyBot at home.

Exclusion criteria:

* Modified Ashworth Scale > 2 for one or more of the following muscles: shoulder adductors, forearm pronator and supinator, flexors and extensors of elbow, wrist and fingers.
* Moderate to severe aphasia: Goodglass-Kaplan's scale < 3.
* Moderate to severe cognitive deficits: levels of cognitive functioning-revised (LCF-R) < 9.
* Functional impairment of the upper limb due to other pathologies.
* Severe pain in the affected arm: visual analogue scale for pain (VASp) ≥ 5.
* Other pathologies which may interfere with the study.
* After discharge, the patient will go to an assisted living facility (e.g., care home).

Eligibility criteria for orthopedic patients

Inclusion criteria:

* Informed Consent signed by the subject.
* Female and male patients between 18 and 90 years old.
* Clinic stay due to an orthopedic-related condition (e.g., surgery, trauma, burns).
* Presence of a motor and/or sensory impairment of the upper limb as assessed by the responsible therapist.
* Possibility (e.g., enough space) to set up the ReHandyBot at home.

Exclusion criteria:

* Moderate to severe aphasia: Goodglass-Kaplan's scale < 3.
* Moderate to severe cognitive deficits: levels of cognitive functioning-revised (LCF-R) < 9.
* Functional impairment of the upper limb due to other pathologies.
* Severe pain in the affected arm: visual analogue scale for pain (VASp) ≥ 5.
* Other pathologies which may interfere with the study.
* After discharge, the patient will go to an assisted living facility (e.g., care home).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose of unsupervised therapy - Minutes | This is measured during the intervention (i.e., during the six weeks of unsupervised therapy at home).
  Dose in minutes of self-administered robot-assisted therapy performed by subjects in the home setting without supervision.
Dose of unsupervised therapy - Repetitions | This is measured during the intervention (i.e., during the six weeks of unsupervised therapy at home).
  Daily dose in number of task repetitions of self-administered robot-assisted therapy performed by subjects in the home setting without supervision.
Dose of unsupervised therapy - Percentual change in therapy time | This is measured during the intervention (i.e., during the six weeks of unsupervised therapy at home).
  Percentage increase in therapy time due to the unsupervised robotic therapy compared to the case where the participants would perform conventional (i.e., normally prescribed) therapy only.

SECONDARY OUTCOMES:
Feasibility - Adverse events | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Feasibility of therapy with the ReHandyBot as assessed by the number of adverse events occurring during this study.
Feasibility - Device deficiencies | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Feasibility of therapy with the ReHandyBot as assessed by the number of device deficiencies occurring during this study.
Feasibility - App deficiencies | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Feasibility of support via RehabCoach as assessed by the number of app deficiencies occurring during this study.
Feasibility - Number of subjects performing unsupervised robot-assisted training | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Feasibility of unsupervised therapy with the ReHandyBot as assessed by the number of subjects who can transition to unsupervised robot-assisted therapy at home out of the total number of tested subjects.
Feasibility - Attendance | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Feasibility of unsupervised therapy with the ReHandyBot as assessed by attendance during the unsupervised phase at home. Attendance is measured as the percentage of days where the subject trains at least once without supervision out of the 42 days offered for unsupervised training at home.
Usability as assessed by the System Usability Scale (1) | This is measured during the intervention (at the end of the familiarization phase, before the 6 weeks unsupervised at home start).
  Usability of the ReHandyBot measured with the System Usability Scale. The possible response options vary between 1 (strongly disagree) and 5 (strongly agree).
Usability as assessed by the System Usability Scale (2) | Usability is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  Usability of the ReHandyBot measured with the System Usability Scale. The possible response options vary between 1 (strongly disagree) and 5 (strongly agree).
Usability as assessed by the raw NASA Task Load Index (1) | This is measured during the intervention (at the end of the familiarization phase, before the 6 weeks unsupervised at home start).
  Usability of the ReHandyBot measured with the raw NASA Task Load Index.
Usability as assessed by the raw NASA Task Load Index (2) | Usability is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  Usability of the ReHandyBot measured with the raw NASA Task Load Index.
Usability as assessed by the mHealth App Usability Questionnaire (MAUQ) for RehabCoach (1) | This is measured during the intervention (at the end of the familiarization phase, before the start of the 6 weeks unsupervised at home).
  Usability of the RehabCoach app measured with the mHealth App Usability Questionnaire (MAUQ). This questionnaire consists of 16 items, with response options ranging from 1 (strongly disagree) to 7 (strongly agree).
Usability as assessed by the mHealth App Usability Questionnaire (MAUQ) for RehabCoach (2) | This is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  Usability of the RehabCoach app measured with the mHealth App Usability Questionnaire (MAUQ). This questionnaire consists of 16 items, with response options ranging from 1 (strongly disagree) to 7 (strongly agree).
Usability as assessed by the Chatbot Usability Questionnaire (1) | This is measured during the intervention (at the end of the familiarization phase, before the start of the 6 weeks unsupervised at home).
  Usability of the RehabCoach chatbots measured with the Chatbot Usability Questionnaire (CUQ). This questionnaire consists of 16 items, with response options ranging from 1 (strongly disagree) to 5 (strongly agree).
Usability as assessed by the Chatbot Usability Questionnaire (2) | This is is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  Usability of the RehabCoach app measured with the Chatbot Usability Questionnaire (CUQ). This questionnaire consists of 16 items, with response options ranging from 1 (strongly disagree) to 5 (strongly agree).
Technology acceptance as assessed by the Technology Acceptance Model | This will be measured at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  Technology acceptance of the RehabCoach app assessed using the Technology Acceptance Model (TAM). This instrument evaluates key constructs such as Perceived Usefulness, Perceived Ease of Use, Attitude Toward Using, and Intention to Use, with responses measured on a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree).
Evolution of patient's satisfaction with robot-assisted therapy as assessed by a 5-point scale | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  A 5-point scale is presented by the robot at the end of each therapy session to measure patient's satisfaction with robot-assisted therapy.
Change in usability metrics between familiarization and end of study | This is calculated at the end of the study (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change in the metrics used to assess usability between the first and second time when they are measured. This change is used to define how the absence of the therapist during robot assisted therapy impacts the perceived usability of the device.
User experience - Customer Satisfaction Score - ReHandyBot (1) | This is measured during the intervention (at the end of the familiarization phase, right before the start of the 6 weeks unsupervised at home).
  The Customer Satisfaction Score consists of the question "Overall, how satisfied are you with the therapy with ReHandyBot?". The possible response options vary between 1 (extremely dissatisfied) and 5 (extremely satisfied).
User experience - Customer Satisfaction Score - ReHandyBot (2) | User experience is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  The Customer Satisfaction Score consists of the question "Overall, how satisfied are you with the therapy with ReHandyBot?". The possible response options vary between 1 (extremely dissatisfied) and 5 (extremely satisfied).
User experience - Net Promoter Score - ReHandyBot (1) | This is measured during the intervention (at the end of the familiarization phase, right before the start of the 6 weeks unsupervised at home).
  The Net Promoter Score consists of the question "How likely would you be to recommend therapy with ReHandyBot to another patient?". The possible response options vary between 1 (extremely unlikely) and 10 (extremely likely).
User experience - Net Promoter Score - ReHandyBot (2) | User experience is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  The Net Promoter Score consists of the question "How likely would you be to recommend therapy with ReHandyBot to another patient?". The possible response options vary between 1 (extremely unlikely) and 10 (extremely likely).
Change in the user experience metrics - ReHandyBot (i.e., Customer Satisfaction Score and Net Promoter Score) | This is calculated at the end of the study (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change in the metrics used to assess user experience for ReHandyBot (i.e., Customer Satisfaction Score and Net Promoter Score) between the first and second time when they are measured. This change is used to define how the absence of the therapist during robot assisted therapy impacts user experience when training with the device.
Reasons for Missing Therapy Sessions | This is calculated at the end of the study (i.e., at the end of the six weeks of unsupervised therapy at home).
  A custom question evaluating the reasons (if any) for not attending the therapy sessions with the device.
User experience - Customer Satisfaction Score - RehabCoach (1) | This is measured during the intervention (at the end of the familiarization phase, right before the start of the 6 weeks unsupervised at home).
  The Customer Satisfaction Score consists of the question "Overall, how satisfied are you with RehabCoach?". The possible response options vary between 1 (extremely dissatisfied) and 5 (extremely satisfied).
User experience - Customer Satisfaction Score - RehabCoach (2) | User experience is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  The Customer Satisfaction Score consists of the question "Overall, how satisfied are you with RehabCoach?". The possible response options vary between 1 (extremely dissatisfied) and 5 (extremely satisfied).
User experience - Net Promoter Score - RehabCoach (1) | This is measured during the intervention (at the end of the familiarization phase, right before the start of the 6 weeks unsupervised at home).
  The Net Promoter Score consists of the question "How likely would you be to recommend RehabCoach to another patient?". The possible response options vary between 1 (extremely unlikely) and 10 (extremely likely).
User experience - Net Promoter Score - RehabCoach (2) | User experience is measured again at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  The Net Promoter Score consists of the question "How likely would you be to recommend RehabCoach to another patient?". The possible response options vary between 1 (extremely unlikely) and 10 (extremely likely).
Change in the user experience metrics - RehabCoach (i.e., Customer Satisfaction Score and Net Promoter Score) | This is calculated at the end of the study (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change in the metrics used to assess user experience with RehabCoach (i.e., Customer Satisfaction Score and Net Promoter Score) between the first and second time when they are measured. This change is used to define how the absence of the therapist during robot assisted therapy impacts user experience when using the RehabCoach app.
Therapeutic alliance as assessed by the Session Alliance Questionnaire | Every day during the 6 weeks unsupervised at home intervention period.
  The Session Alliance Questionnaire (SAQ), administered through the chatbot throughout the intervention, to measure therapeutic alliance at the session level.
Smartphone usage and familiarity with texting apps as assessed by two custom questions | This is assessed after the familiarization period, before the 6-weeks intervention starts.
  Custom questions assessing participants' general smartphone usage frequency (ranging from "never" to "more than 2 hours per day") and familiarity with texting applications (e.g., WhatsApp), ranging from "not familiar" to "very familiar." These questions provide contextual information on participants' baseline technology use.
Qualitative analysis of conversational data with RehabCoach chatbots | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  A qualitative analysis of the conversational data collected by RehabCoach to evaluate interaction patterns and patient engagement. This will be used to evaluate which conversations contributed to users adherence to ReHandyBot therapy.
Educational material knowledge retention as assessed by quiz performance | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  The feasibility and effectiveness of the educational program delivered by RehabCoach will be assessed through the number of correct answers on quizzes administered immediately after each educational topic.
Engagement as assessed by number of educational sessions completed | Recorded throughout the intervention period, measured at the end of the 6-weeks intervention.
  Engagement with the educational program will be assessed by recording the number of sessions patients complete within the RehabCoach app.
Motivation as assessed by therapy session adherence and initiation | Measured at the end of the study protocol (i.e., at the end of the six weeks of unsupervised therapy at home).
  The impact of RehabCoach on motivation to train with ReHandyBot will be determined by (1) the number of unscheduled or additional therapy sessions initiated by patients beyond the minimum daily recommendation, and (2) the comparison between the number of sessions scheduled with RehabCoach and the number of sessions actually performed.
Change in upper limb functions as assessed by the ABILHAND | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the ABILHAND scale.
Change in upper limb functions as assessed by the Box and Block (BBT) test | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) upper limb functions as assessed by the BBT test.
Change in Upper Limb Function as Assessed by the Box and Block Test (BBT) | Measured at baseline and at the end of the study protocol (after six weeks of unsupervised therapy at home).
  Change in upper limb function will be assessed using the Box and Block Test (BBT). Performance will be compared between baseline (beginning of the study) and post-intervention (end of the study).
Change in Sensory Function as Assessed by the Erasmus MC Modification to the Revised Nottingham Sensory Assessment (EmNSA) | Measured at baseline and at the end of the study protocol (after six weeks of unsupervised therapy at home).
  Change in sensory function will be assessed using the Erasmus MC modification to the revised Nottingham Sensory Assessment (EmNSA), which evaluates tactile sensation, proprioception, and stereognosis. Performance will be compared between baseline (beginning of the study) and post-intervention (end of the study).
Change in the active Range of Motion (aROM) for grasping measured in millimeters as assessed by the custom robotic assessment "aROM - Hand" | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) aROM for grasping, i.e. for hand opening and closing. This is measured by the robot with a custom assessment.
Change in the active Range of Motion (aROM) for forearm rotation measured in degrees as assessed by the custom robotic assessment "aROM - Forearm" | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) aROM for forearm pronation and supination. This is measured by the robot with a custom assessment.
Change in proprioception as assessed by the custom robotic assessment "JND" measuring the minimum difference in length (mm) and/or angle (degrees) that a patient can perceive | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) proprioception, defined as the minimum difference in length and/or angle that a patient can perceive (i.e. just noticeable difference). This is measured by the robot with a custom assessment.
Change in haptic perception as assessed by the custom robotic assessment "Weber Fraction" measuring the minimum difference in stiffness that a patient can perceive in percentage | This is calculated at the end of the study, after performing the final measurements (i.e., at the end of the six weeks of unsupervised therapy at home).
  Change between baseline (i.e. beginning of the study) and final (i.e. end of the study) haptic perception, defined as the minimum difference in stiffness that a patient can perceive expressed in percentage according to the Weber Fraction law . This is measured by the robot with a custom assessment named "Weber fraction".
Content of robotic therapy - Intensity | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Intensity (i.e., repetitions over time) of the robotic therapy throughout the study.
Content of robotic therapy - Performance | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Task performance (i.e., correct trials over total trials) during robotic therapy throughout the study.
Content of robotic therapy - Effective time ratio | This is monitored over the whole protocol duration (i.e., from beginning of the first week to the end of the six weeks of unsupervised therapy at home).
  Ratio of effective (i.e., net total therapy time without breaks) over total duration of the therapy session during robotic therapy throughout the study.
Parameters influencing unsupervised robot-assisted therapy | This is calculated at the end of the study (i.e., at the end of the six weeks of unsupervised therapy at home).
  Correlation between achieved unsupervised robot-assisted therapy dose and different parameters (i.e., cognitive assessments (Goodglass-Kaplan Scale, LCF-R, Montreal Cognitive Assessment (MoCA)) performed during the screening visit, the clinical assessments, the robotic assessments, demographics and the collected medical data).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lambercy, Prof. Dr., Principal Investigator — Swiss Federal Institute of Technology Zurich

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy considerations and because the dataset will not be large enough to support meaningful secondary analyses.

REFERENCES:
- [Background] Devittori, G., Akeddar, M., Retevoi, A., Schneider, F., Cvetkova, V., Dinacci, D., Califfi, A., Rossi, P., Petrillo, C., Kowatsch, T., & Lambercy, O. (2024). Towards RehabCoach: Design and Preliminary Evaluation of a Conversational Agent Supporting Unsupervised Therapy After Stroke. 2024 10th IEEE RAS/EMBS International Conference for Biomedical Robotics and Biomechatronics (BioRob), 569-574. https://doi.org/10.1109/BIOROB60516.2024.10719881